CLINICAL TRIAL: NCT04820673
Title: A Real-world Prospective Cohort Study of Patients With Moderate to Severe Acne Vulgaris Treated With Sarecycline (Seysara®) In Community Practice Settings in the U.S
Brief Title: Patient-reported Outcomes for Sarecycline Effectiveness and Safety (PROSES)
Acronym: PROSES
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: M-24001-40
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Acne Vulgaris
Keywords: Prospective; Non-nodular Acne Vulgaris; Perceptions; Health-Related Quality of Life (HRQoL); Patient-Reported Outcomes (PROs); Signs & Symptoms
MeSH Terms: conditions — Acne Vulgaris; Signs and Symptoms | interventions — sarecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sarecycline: Eligible patients prescribed with commercially available sarecycline will be followed-up for 12 weeks post-initiation of treatment.
  Interventions: Drug: Sarecycline

INTERVENTIONS:
Drug: Sarecycline — Clinicians will prescribe the sarecycline as per their own clinical judgment and standard practice.
  Other Names: Seysara®

SUMMARY:
The purpose of this study is to evaluate the patient-reported outcomes (PROs) in terms of health-related quality of life (HRQoL) and signs of Acne Vulgaris (AV) among patients with moderate to severe non-nodular AV who are administered sarecycline (Seysara®) in real-world community practice settings in the United States (U.S). Investigator's Global Assessment (IGA) of AV and safety measures associated with use of sarecycline (Seysara®) will be assessed over the study observation period of 12 weeks. Clinicians will prescribe sarecycline (Seyara®) as per their own clinical judgment and standard practice.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* Male or female, aged 9 years and above
* Has facial non-nodular AV with IGA score of moderate or severe
* Considered as a potential candidate for sarecycline (Seysara®) treatment, per clinician judgment

Caregiver Inclusion Criteria:

* Primary caregiver of the study-eligible patient
* Male or female, aged 18 years and above

Exclusion Criteria:

* Patients with any known resistance to other tetracyclines
* Patients with any dermatological or physical condition of the face that could interfere with the AV clinical evaluations.
* Patients with any history of allergy to tetracycline-class antibiotics, pseudomembranous colitis or antibiotic-associated colitis.
* Unable to comply with the requirements of the study or patients who in the opinion of the Site Investigator should not participate in the study

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe non-nodular acne vulgaris who are on prescribed sarecycline will be enrolled. Caregivers of eligible pediatric patients will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (2):
- United States (2):
  - Almirall Site#2, Boston, Massachusetts
  - Almirall Site #1, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 30 investigative sites from 09 March 2021 to 04 May 2022.
Pre-assignment Details: A total of 300 Acne Vulgaris (AV) participants were enrolled and received treatment in this study.
Groups:
- Sarecycline: Participants prescribed with commercially available sarecycline 1.5 milligram per kilogram per day (mg/kg/day), tablets, orally were followed for up for 12 weeks post-initiation of treatment.
Period: Overall Study
Arm/Group | Sarecycline
Started | 300
Safety Analysis Set (Safety analysis set included all participants who started the study and received at least one dose of the sarecycline during the study observation period, as part of usual care.) | 300
Full Analysis Set (FAS) (FAS included all participants within the safety population that had at least one question answered pertaining to study primary research objective and who completed their Week-12 survey.) | 253
Completed | 262
Not Completed | 38
Not completed — Adverse Event | 6
Not completed — Due to Lack of Effectiveness | 1
Not completed — Pregnancy | 1
Not completed — Voluntary Withdrawal | 20
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of sarecycline during the study observation period, as part of usual care.
Groups:
- Sarecycline: Participants prescribed with commercially available sarecycline 1.5 mg/kg/day, tablets, orally were followed for up for 12 weeks post-initiation of treatment.
Arm/Group | Sarecycline
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116
  Between 18 and 65 years | 184
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic, Latino, or of Spanish Origin | 101
  Ethnicity: Other | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 195
  Race: Black or African American | 32
  Race: American Indian or Alaska Native | 3
  Race: Asian | 17
  Race: Native Hawaiian or Other Pacific Islander | 3
  Race: Other | 41
  Race: Prefer not to answer | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Acne Symptom and Impact Scale Questionnaire (ASIS) Domain Score at Week 12
Description: Patient related outcome (PROs) assessment performed using ASIS Questionnaire, a 17-item questionnaire that asks participants about the signs, impact (emotional and social) of AV, responses were reported as two scales: Signs (9 items), and Impact (8 items). Impact domain had two sub-scales, pertinent to Emotional (6 items) and Social impact (2 items). All items are scored on a 5-point scale: 0 (best) to 4 (worst). A domain score is determined by the average of scores in each scale within the domain. The total score is the average of all 17 items. Higher scores on the ASIS Sign domain, comprised of all items that assess symptoms (items 1-9), indicate the presence of more severe symptoms, whereas higher scores on the ASIS Impact domain, comprised of all the items that assess impacts (items 10-17), indicate a greater negative impact of acne.
Time Frame: Baseline, Week 12
Population: FAS included all participants within the safety population that had at least one question answered pertaining to study primary research objective and who completed their Week-12 survey.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Sarecycline
Number analyzed (Participants) | 253
Score on a Scale
  Signs Domain Score: Baseline | 1.96 (0.58)
  Signs Domain Score: Change at Week 12 | -0.77 (0.67)
  Impact Domain Score: Baseline | 2.06 (0.91)
  Impact Domain Score: Change at Week 12 | -1.01 (1.03)
  Emotional Impact Domain Score: Baseline | 2.43 (0.96)
  Emotional Impact Domain Score: Change at Week 12 | -1.15 (1.12)
  Social Impact Domain Score: Baseline | 0.98 (0.99)
  Social Impact Domain Score: Change at Week 12 | -0.60 (1.06)
Statistical Analysis 1: Comparison: Sarecycline; Week 12 vs Baseline; Test type: Other; p < .0001, t-test, 2 sided — P<0.0001, calculated by t-test, corresponds to baseline response group domain scores in comparison to week-12 domain scores (CFB). CFB is calculated using available matching data for each domain. Higher domain scores indicate higher disease burden

2. Secondary Outcome: Percentage of Participants With Facial Investigator Global Assesment (IGA) Success at Week 12
Description: The investigator assessed the participant's facial acne using the IGA 5-point scale. The scale ranges from 0 (best): clear, no evidence of papules or pustules to 4 (worst): severe, inflammatory lesions are more apparent, many papules/pustules, there may or may not be a few nodulocytic lesions. Success was defined as at least a 2-point decrease (improvement) from Baseline on the IGA assessment as well as a score of clear (0) or almost clear (1). Percentage of participants who achieved facial IGA success at Week 12 were reported.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sarecycline
Number analyzed (Participants) | 253
Percentage of Participants | 58.89

ADVERSE EVENTS:
Time Frame: From start of study up to Week 12
Description: Safety analysis set included all participants who started the study and received at least one dose of the sarecycline during the study observation period, as part of usual care.
Arm/Group | Sarecycline
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 1/300
Other Adverse Events (participants affected / at risk) | 30/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarecycline (N=300)
Idiopathic intracranial hypertension (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarecycline (N=300)
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (upper) (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Injury associated with device (General disorders) | 1
COVID-19 (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2
Animal bite (Injury, poisoning and procedural complications) | 1
Weight Increased (Investigations) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 2
Migraine with aura (Nervous system disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04820673/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT04820673/SAP_001.pdf